CLINICAL TRIAL: NCT01945736
Title: Pharmacokinetics of Multiple Dose Methadone in Children
Brief Title: Pharmacokinetics of Multiple Dose Methadone in Children Treated for Opiate Withdrawal
Acronym: MTH01
Status: Completed | Type: Observational
Sponsor: Kevin Watt (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Kevin Watt, Assistant Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00044082; HHSN27500021 (Other: NICHD)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Opiate Withdrawal Syndrome
Keywords: Opiate withdrawal in children
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The Study team is interested in learning more about how genetic differences in proteins known as cytochrome P450 enzymes effect the breakdown of methadone. The study team will gather leftover blood collected from the infant or child while the infant/child was in this study and send it to a laboratory to test for genetics. There will be no extra blood draws for this part of the study.
  The samples for genetic testing will be given a code number and will not be labeled with the infant or child's name or initials, or any other information that could identify the infant or child. Any remaining blood will be destroyed after the genetic laboratory testing is complete.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cohort 1: > or = 90 days to < 2 years on enteral methadone. Dose schedule is per routine medical care.
  Interventions: Drug: Methadone
- Cohort 2: 2 years to < 6 years on enteral methadone. Dose schedule is per routine medical care. Will include overweight children with BMI for age of 85 - 95 percentile, or obese children BMI for age > or = to 95 percentile.
  Interventions: Drug: Methadone
- Cohort 3: 6 years to < 18 years on enteral methadone. Dose schedule is per routine medical care. Will include overweight children with BMI for age of 85 - 95 percentile, or obese children BMI for age > or = to 95 percentile.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — To determine the PK of enteral methadone in children > or = 90 days and <18 years treated for opiate withdrawal per routine medical care.

SUMMARY:
The purpose of this study is to learn more about how the study drug, methadone, prescribed by an infant's or child's physician as part of standard medical care, is processed in children and young adults. While this drug is used extensively in infants and children, it has not been extensively studied in this population.

Physicians do not have very much information on how long it takes for methadone to be removed from the blood circulation and passed out of the body. Physicians need more information to guide how much and how often we should give methadone to children/young adults to ensure they get the maximum effect with the minimum amount of drug. During this research study, the study team will collect information about how this drug is processed in infants and children.

DETAILED DESCRIPTION:
A total of approximately 24 to 36 infants and children will participate in this study. This study will be done at five medical centers in the United States.

Treatment will be prescribed by the infant or child's doctor and not by the study team.

Participants will be divided into 3 groups based on age, ages 3 months to 2 years, ages 2 to 6 years, and ages 6 to 18 years. There will be approximately 8 to 12 participants enrolled in each group. Additionally, at least 6 overweight or obese participants between ages 2-18 years will be included in this study.

Information collected from each subject's routine medical care will include:

* Participant gender, date of birth, race and ethnicity
* Pertinent medical history
* Laboratory results (blood count and chemistries) from routine testing ordered by the infant or child's regular doctor
* Medications of interest the child was given within the 72 hours prior to first dose of methadone administered after consent
* Time and dose of methadone administered to the child up to 14 days prior to enrollment

Study specific information collected will include:

* Blood sample collection to measure level of methadone
* Baseline WAT-1 score (sedation withdrawal assessment of the infant or child used to assess symptoms the child/infant may experience when opioid drugs are discontinued).

The duration of the study will be up to 10 days, comprised of a maximum 5 day treatment period a 5 day observation period.

ELIGIBILITY:
Inclusion Criteria:

* >90 days - < 18 years of age at the time of first dose of study drug
* Receiving enteral methadone as standard of care
* Signed informed consent/HIPAA documents by the parent/legal guardian and assent (if applicable)

Exclusion Criteria:

* Previous participation in the study
* Subject is receiving ECLS (Extracorporeal Life Support)
* < 36 weeks gestational age at birth for children <1 year of age at time of enrollment
* Any other condition or chronic illness that in the opinion of the Principal
* Investigator makes participation unadvised or unsafe

Ages: 91 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be divided into 3 groups based on age, ages 3 months to 2 years, ages 2 to 6 years, and ages 6 to 18 years. There will be approximately 8 to 12 participants enrolled in each group. Additionally, at least 6 overweight or obese participants between ages 2-18 years will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
PK Parameters after multiple doses of enteral methadone | Maximum of 7 PK samples based on dosing schedule collected over a 5 day period
  * Apparent oral clearance
  * Apparent oral volume of distribution
  * Area under the curve
  * Absorption rate constant

SECONDARY OUTCOMES:
PK of methadone's primary metabolite EDDP | Maximum of 7 PK samples based on dosing schedule collected over a 5 day period
PK of R- and S-enantiomers of methadone | Maximum of 7 PK samples based on dosing schedule collectes over a 5 day period
Correlation between plasma and DBS samples | Maximum of 7 PK samples based on dosing schedule collected over a 5 day period
Correlation between plasma and scavenge samples | Maximum of 7 PK samples based on dosing schedule collected over a 5 day period
Influence of CYP3A4 and CYP3B6 genetic polymorphisms on methadone PK | Maximum of 7 PK samples based on dosing schedule collected over a 5 day period
Methadone pharmacodynamics using the WAT-1 | Maximum of 7 PK samples based on dosing schedule collected over a 5 day period
Adverse events | Study days 1-5 and observational days 6-10

CONTACTS AND LOCATIONS:
Overall Officials: Kevin watt, MD, Principal Investigator — Duke Medical Center/Duke Clinical Research Institute
Locations (5):
- United States (5):
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Mercy Hospital, Kansas City, Kansas
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina